CLINICAL TRIAL: NCT01789476
Title: A Single-Center, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Analgesic Efficacy and Safety of CR845 Dosed in Patients With Pain Following Bunionectomy Surgery
Brief Title: A Phase 2 Study to Evaluate Analgesic Effect of IV CR845 For Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR845 CLIN2003
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Acute Pain
Keywords: pain; acute pain; kappa agonis; opioid analgesia; bunionectomy; peripheral nervous system agents; physiological effects of drugs; surgery; post-operative; post-operative complications
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR845 (Experimental): Peripheral kappa opioid receptor agonist
  Interventions: Drug: CR845
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 — CR845 dosage = 0.005 mg/kg per dose, IV bolus. The initial dose was administered upon reaching a qualifying pain intensity score and followed by a supplemental dose, if requested by patient for pain. Additional doses could be administered every 8 hours up to 48 hours.
  Other Names: Active treatment for post-operative pain
  Arms: CR845
Drug: Placebo — Matching placebo administered using same dosing algorithm as the active arm
  Other Names: Post-operative placebo for pain
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double blind, placebo controlled, parallel group proof of concept study to evaluate the analgesic efficacy as well as the safety, tolerability and pharmacokinetic profile of CR845 in patients with pain following bunionectomy surgery.

DETAILED DESCRIPTION:
Currently, the most widely used drugs to treat pain after surgery are opiates, such as morphine. Morphine works mainly by activating one of several types of opiate receptors that control some of our pain sensation - the so-called mu opiate receptors. These receptors are located in many areas of the brain and also outside of the brain. By activating these receptors, morphine provides significant pain relief, but also causes side effects that limit its use. Some of these side effects include: respiratory depression or arrest (slowed or stopped breathing), sedation (a state of calmness or extreme relaxation), euphoria (an exaggerated feeling of physical and mental well-being), constipation, nausea, vomiting, and drug addiction.

In order to avoid the side effects of morphine and other mu opiates, the present experimental drug CR845 was designed to work at a different type of opiate receptor - called kappa - that can also provide pain relief, by acting on sensory nerves outside the brain. CR845 was designed to penetrate the brain much less than other opiate drugs, which should result in pain relief similar to that of morphine, but with fewer side effects. Because CR845 activates kappa receptors instead of mu receptors, the side effects are different than with a morphine-type drug. In particular, kappa opiates, such as CR845, do not cause respiratory depression or arrest, euphoria, constipation, drug tolerance, physical drug dependence or drug addiction. For these reasons, CR845 may present a distinct advantage over other opiates that are currently used for pain relief and post-operative pain in particular.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to any study procedures;
2. Able to communicate clearly with the Investigator and staff;
3. Males and females aged 18 years or older;
4. Scheduled for elective primary unilateral first metatarsal bunionectomy surgery (osteotomy and internal fixation) with no collateral procedures;
5. Females physically incapable of childbearing potential (postmenopausal for more than 1 year or surgically sterile) or practicing an acceptable method of contraception (hormonal, barrier with spermicide, intrauterine device, vasectomized partner, or abstinence). Subjects using hormonal birth control must have received at least 1 cycle of treatment prior to randomization. All females of childbearing potential must have a negative pregnancy test and not be breast feeding at Baseline;
6. Negative urine drug screen for drugs of abuse at Screening and at Baseline; a positive drug screen result may be permitted if the patient has been on a stable dose of an allowed medication for >30 days (antipsychotics, antiepileptics, sedatives, hypnotics, or antianxiety agents, selective serotonin reuptake inhibitors [SSRIs], tricyclic antidepressants) or >3 months (opioid analgesics or systemic steroids);
7. American Society of Anesthesiologists (ASA) risk class of I to II;
8. Body weight <170 kg

Exclusion Criteria:

1. Has known allergies to opioids, unless has subsequently tolerated other opioids and in the opinion of the PI could tolerate study drug;
2. Has a known or suspected history of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)-diagnosed alcohol, opiate or other drug abuse or dependence within 12 months prior to screening;
3. Is unable to refrain from alcohol consumption for a period beginning 24 hours prior to surgery through the end of the Treatment Period;
4. Has taken non-opioid analgesics (including cyclooxygenase-2 [COX-2] inhibitors) or nonsteroidal anti-inflammatory drugs (NSAIDs) within 12 hours of the Baseline assessments;
5. Has taken any opioid analgesics or used systemic steroids within 4 days of surgery OR has been using opiates chronically for a period of < 3 months; (Note: Patients on stable chronic opioids for ≥ 3 months will need to discontinue them for 4 days prior to surgery);
6. Has used antipsychotics, antiepileptics, sedatives, hypnotics, or antianxiety agents, selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants for < 30 days prior to surgery or had a dose change within the previous 30 days;
7. Has taken any prescription or over-the-counter medication within 4 days prior to surgery that, in the opinion of the Investigator, is expected to confound the analgesic response;
8. Has taken herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) during any of the 7 days prior to surgery;
9. Has any clinically significant condition or a significant laboratory abnormality that would, in the Investigator's or designee's opinion, preclude study participation
10. Has received another investigational drug within 30 days of scheduled surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Muse, MD, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CR845: CR845 (0.005 mg/kg) IV
Period: Overall Study
Arm/Group | CR845 | Placebo
Started | 34 | 17
Completed | 26 | 15
Not Completed | 8 | 2
Not completed — Lack of Efficacy | 6 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Unable to get IV access | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | CR845 | Placebo | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 16 | 48
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 16 | 45
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 29 | 17 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 32 | 15 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Differences Over 24 Hours (SPID 0-24) Following the Initial Administration of Study Drug
Description: Patients reported their pain intensity using a visual analogue scale (VAS) from 0 to 100 mm, where 0 mm represented "No Pain" and 100 mm represented the "Worst Pain You Can Imagine". SPID 0-24 represents the cumulative time-weighted sum of the pain intensity difference (PID) scores between each assessment timepoint following the postoperative administration of study drug (i.e. 0 to 15 min, 15 to 30 min, etc.) over 24 hours. Pain intensity assessments were measured at baseline (entry pain score) and at 15, 30, 45, 60, 90, 120 and 150 minutes; 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 hours after the first administration of study drug (only timepoints up to 24 hours used in calculating SPID 0-24).
  Negative SPID values represent a decrease in pain intensity (i.e. lower values indicate a greater reduction in pain).
Time Frame: 0 to 24 hours
Population: The analysis included all patients in the Completer population who completed the trial, where time 0 was the start time of the first dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 15 | 26
units on a scale * hours | -52.08 (395.02) | -292.7 (390.52)
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p < 0.05, ANOVA — One-sided ANOVA with Treatment Group as a Main Effect

2. Secondary Outcome: Summed Pain Intensity Differences Over 36 Hours (SPID 0-36) Following the Initial Administration of Study Drug
Description: Patients reported their pain intensity using a visual analogue scale (VAS) from 0 to 100 mm, where 0 mm represented "No Pain" and 100 mm represented the "Worst Pain You Can Imagine". SPID 0-24 represents the cumulative time-weighted sum of the pain intensity difference (PID) scores between each assessment timepoint following the postoperative administration of study drug (i.e. 0 to 15 min, 15 to 30 min, etc.) over 24 hours. Pain intensity assessments were measured at baseline (entry pain score) and at 15, 30, 45, 60, 90, 120 and 150 minutes; 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 hours after the first administration of study drug (only timepoints up to 36 hours used in calculating SPID 0-36).
  Negative SPID values represent a decrease in pain intensity (i.e. lower values indicate a greater reduction in pain).
Time Frame: Up to 36 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 15 | 26
units on a scale * hours | -259.2 (533.24) | -675.6 (658.0)
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p < 0.03, ANOVA — One-sided ANOVA with Treatment Group as a Main Effect

3. Secondary Outcome: Summed Pain Intensity Differences Over 48 Hours (SPID 0-48) Following the Initial Administration of Study Drug
Description: Patients reported their pain intensity using a visual analogue scale (VAS) from 0 to 100 mm, where 0 mm represented "No Pain" and 100 mm represented the "Worst Pain You Can Imagine". SPID 0-24 represents the cumulative time-weighted sum of the pain intensity difference (PID) scores between each assessment timepoint following the postoperative administration of study drug (i.e. 0 to 15 min, 15 to 30 min, etc.) over 24 hours. Pain intensity assessments were measured at baseline (entry pain score) and at 15, 30, 45, 60, 90, 120 and 150 minutes; 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 hours after the first administration of study drug.
  Negative SPID values represent a decrease in pain intensity (i.e. lower values indicate a greater reduction in pain).
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 15 | 26
units on a scale * hours | -534.4 (724.8) | -1117 (954.8)
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p < 0.03, ANOVA — One-sided ANOVA with Treatment Group as a Main Effect

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the start of study drug administration to the Follow-up visit (up to Day 10 after surgery).
Arm/Group | CR845 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 29/34 | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR845 (N=34) | Placebo (N=17)
Dizziness (Nervous system disorders) | 10 (10) | 4 (4)
Paraesthesia (Nervous system disorders) | 10 (13) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 10 (13)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infusion site bruising (General disorders) | 2 (2) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 1 (1)
Injection site discharge (General disorders) | 1 (1) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days